CLINICAL TRIAL: NCT04823923
Title: Study of the Impact of the Stage of Chronic Renal Failure on Plasma Exposure of Kinase Inhibitors (ITK) in Patients Treated for Metastatic Kidney Cancer
Brief Title: Impact of Chronic Renal Failure on Plasma Exposure of Kinase Inhibitors in Patients Treated for Metastatic Kidney Cancer
Acronym: IREKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROICM 2020-08 IRE; 2020-A01533-36 (Other: ID RCB number of competent autority in France)
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Kidney Neoplasm
Keywords: metastatic kidney cancer; pazopanib; cabozantinib; renal failure
MeSH Terms: conditions — Kidney Neoplasms; Renal Insufficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Patients without renal insufficiency under pazopanib (Other): Pazopanib is taken daily, for a minimum of 3 months, according to the medical prescription.
  Interventions: Other: blood sampling for ITK dosage
- Patients without renal insufficiency under cabozantinib (Other): Cabozantinib is taken daily, for a minimum of 3 months, according to the medical prescription.
  Interventions: Other: blood sampling for ITK dosage
- Patients with moderate renal impairment under pazopanib (Other): Pazopanib is taken daily, for a minimum of 3 months, according to the medical prescription.
  Interventions: Other: blood sampling for ITK dosage
- Patients with moderate renal impairment under cabozantinib (Other): Cabozantinib is taken daily, for a minimum of 3 months, according to the medical prescription.
  Interventions: Other: blood sampling for ITK dosage
- Patients with severe or terminal stage renal impairment under pazopanib (Other): Pazopanib is taken daily, for a minimum of 3 months, according to the medical prescription.
  Interventions: Other: blood sampling for ITK dosage
- Patients with severe or terminal stage renal impairment under cabozantinib (Other): Cabozantinib is taken daily, for a minimum of 3 months, according to the medical prescription.
  Interventions: Other: blood sampling for ITK dosage

INTERVENTIONS:
Other: blood sampling for ITK dosage — Blood sample for ITK dosage at visit 1 (1 month +/- 1 week after the start of treatment) and at visit 2 (3 months +/- 1 month after the start of treatment)

SUMMARY:
The study of the blood concentration of ITK what are pazopanib and cabozantinib at 1 month and 3 months from the start of treatment will allow to evaluate the impact of renal failure on their efficacy and toxicity in patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
This study involves patients treated with cabozantinib or pazopanib in their metastatic renal cancer.

Indeed, the aim of this study is to assess the blood concentration of these two drugs as well as their tolerance, in relation to their renal function (normal renal function or moderate or severe renal failure).

Pazopanib and cabozantinib are kinase inhibitors that are indicated for a number of cancer conditions, including metastatic kidney cancer.

Both of these oral therapies require a daily intake of the drug to ensure its effectiveness.

For this, the patient must have optimal compliance and benefit from regular follow up to assess clinical and biological tolerance.

Chronic renal failure is a factor that may impact the efficacy and toxicity of pazopanib and cabozantinib. This may be due either to a elimination default of the drug or to much elimination if the drug is filtered after dialysis.

As a result, kinase inhibitors could be impacted by chronic renal failure and thus modify the safety and efficacy of the treatment.

A study-specific blood test will be taken at 1 month and at 3 months during a consultation (this blood test is in addition to the routine blood test). Its analysis will evaluate the quantity of medication present in the blood.

The other objective of this study is to evaluate the side effects of the drug taken by the patient (pazopanib or cabozantinib).

This will alow to propose possible dose adjustments for each of these treatments and thus improve the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient followed for metastatic clear cell renal cell carcinoma.
2. Age ≥18 years old.
3. Performance Status (PS) according to Eastern Cooperative Oncology Group (ECOG) = 0, 1 or 2
4. Patient treated with a VEGF-R inhibitor: pazopanib or cabozantinib for metastatic kidney cancer.
5. If patient doesn't have renal failure -> group 1, or if patient has chronic renal failure according to the moderate stage Chronic Kidney Disease - Epidemiology (CKD-EPI) formula (Clr <60 ml / min, stage 3) -> group 2, or if patient have chronic renal failure according to the CKD-EPI formula of severe or terminal stage (Clr <30 ml / min, stage 4 and stage 5), with or without dialysis -> group 3.
6. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
7. Patient having given informed, written and express consent.
8. Affiliation to the French Social Security System.

Exclusion Criteria:

1. Indication other than clear cell renal cell carcinoma for these same ITKs
2. Pregnant or breast-feeding subjects
3. Patient whose regular follow-up is impossible for psychological, family, social or geographic reasons,
4. Patient under guardianship, curatorship or safeguard of justice
5. Participation in another clinical study with a research product during the last 30 days before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Residual concentration at equilibrium of ITK in the blood | at 1 month (+/1 week)
  Assessment in patients treated for metastatic kidney cancer without or with moderate or severe renal impairment if the plasma concentration (residual concentration at equilibrium) of ITK is higher than the target concentration (specific to the ITK molecule : pazopanib : 20 000 ng/mL and cabozantinib : 1000 ng/mL )

SECONDARY OUTCOMES:
Concentration of ITK in the blood in patients with Failure renal function | at 1 month (+/- 1 week) and 3 months (+/- 1 month)
  Assessment the plasma concentration (residual concentration at equilibrium) of ITK (pazopanib and / or cabozantinib) in patients with moderate renal impairment and / or severe renal impairment
Concentration of ITK in the blood in patients with normal renal function | at 1 month (+/- 1 week) and 3 months (+/- 1 month)
  Assessment the plasma concentration (residual concentration at equilibrium) of ITK (pazopanib and / or cabozantinib) in patients with normal renal function
Toxicities related to the intake of ITKs | at 1 month (+/- 1 week) and 3 months (+/- 1 month)
  Assessment toxicities induced by the use of ITK targeting Vascular Endothelial Growth Factor-Receptor (VEGF-R) by using the NCI-CTCAE version 5.0 (grade ≥ 2)

CONTACTS AND LOCATIONS:
Overall Officials: Fanny LEENHARDT, Dr, Principal Investigator — Institut du Cancer de Montpellier (ICM)
Locations (5):
- France (5):
  - APHM Hôpital LA TIMONE, Marseille
  - CHU Montpellier - Hôpital St Eloi, Montpellier
  - ICM Val d'Aurelle, Montpellier
  - CHU de Nîmes, Institut de Cancérologie du Gard, Nîmes
  - Institut Universitaire du Cancer de Toulouse (IUCT) Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Background] van Erp NP, Gelderblom H, Guchelaar HJ. Clinical pharmacokinetics of tyrosine kinase inhibitors. Cancer Treat Rev. 2009 Dec;35(8):692-706. doi: 10.1016/j.ctrv.2009.08.004. Epub 2009 Sep 5. PMID 19733976
- [Background] Hendrayana T, Wilmer A, Kurth V, Schmidt-Wolf IG, Jaehde U. Anticancer Dose Adjustment for Patients with Renal and Hepatic Dysfunction: From Scientific Evidence to Clinical Application. Sci Pharm. 2017 Feb 27;85(1):8. doi: 10.3390/scipharm85010008. PMID 28264440
- [Background] Verheijen RB, Bins S, Mathijssen RH, Lolkema MP, van Doorn L, Schellens JH, Beijnen JH, Langenberg MH, Huitema AD, Steeghs N; Dutch Pharmacology Oncology Group. Individualized Pazopanib Dosing: A Prospective Feasibility Study in Cancer Patients. Clin Cancer Res. 2016 Dec 1;22(23):5738-5746. doi: 10.1158/1078-0432.CCR-16-1255. Epub 2016 Jul 28. PMID 27470967
- [Background] Lacy S, Yang B, Nielsen J, Miles D, Nguyen L, Hutmacher M. A population pharmacokinetic model of cabozantinib in healthy volunteers and patients with various cancer types. Cancer Chemother Pharmacol. 2018 Jun;81(6):1071-1082. doi: 10.1007/s00280-018-3581-0. Epub 2018 Apr 23. PMID 29687244